CLINICAL TRIAL: NCT04826848
Title: The Prognostic Value of Lactate Clearance in Hospital-acquired Pneumonia
Brief Title: Lactate Clearance in Hospital-acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: LC-HAP
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-03

CONDITIONS: Pneumonia; Mortality; Lactate; Prognosis
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lactate — We will evauate the lactate clearance of the patients in 6 hours period. Lactate clearance = [(Initial lactate - 6th hour lactate) / Initial lactate] * 100

SUMMARY:
There is no clear consensus on the use of pneumonia severity index (PSI) developed for community-acquired pneumonia in hospital-acquired pneumonia cases. In another aspect, PSI is a relatively difficult scoring system that includes many parameters. This study evaluated whether lactate clearance could be used as a mortality marker instead of PSI in hospital-acquired pneumonia. As a result, lactate clearance was lower in the mortal group and when the diagnostic statistics were evaluated, it was seen that the sensitivity and specificity rates were significantly higher. In conclusion, lactate clearance has been evaluated as a strong predictor of mortality in hospital-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over age, hospital-acquired pneumonia, emergency department admissions

Exclusion Criteria:

* Patients who are pregnant or lactating, under 18 years of age, in the healthcare-associated pneumonia group, had mechanical ventilation at the last hospitalization, whose lactate level could not be studied for any reason at admission and 6th hour, had missing data used in pneumonia severity index calculation and/or who did not accept to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the age of 18 and over with at least 48 hours of hospitalization within the specified study date range, who were discharged from the hospital within the last 14 days related to this hospitalization, who were re-admitted to the adult emergency department and were diagnosed with pneumonia were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 day
  28-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alp Şener, MD, Principal Investigator — Ankara Yıldırım Beyazıt University Faculty of Medicine
Locations (1):
- Ankara Yıldırım Beyazıt University, School of Medicine, Department of Emergency Medicine, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No